CLINICAL TRIAL: NCT03774368
Title: Targeted Video Messaging About Emergency Contraception Via a Social Media Platform
Brief Title: Targeted Video Messaging About Emergency Contraception
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Planned Parenthood League of Massachusetts (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2018P001764
Record Dates: First submitted 2018-12-11; First posted 2018-12-13 (Actual); Last update posted 2019-07-16 (Actual); Status verified 2019-07

CONDITIONS: Contraception

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Website about emergency contraception (Other): Subjects are randomly assigned to view an existing website about emergency contraception. The website contains information about the three methods of emergency contraception: the copper IUD, ulipristal pill, and levonorgestrel pill. It includes information about their relative effectiveness and where to access emergency contraception.
  Interventions: Other: Emergency contraception website
- Video about emergency contraception (Other): Subjects are randomly assigned to view an existing video about emergency contraception. The video is two minutes in length and contains information about the three methods of emergency contraception: the copper IUD, ulipristal pill, and levonorgestrel pill. It includes information about their relative effectiveness and where to access emergency contraception.
  Interventions: Other: Emergency contraception video

INTERVENTIONS:
Other: Emergency contraception website — Existing website with factual information about emergency contraception
  Arms: Website about emergency contraception
Other: Emergency contraception video — Existing video with factual information about emergency contraception
  Arms: Video about emergency contraception

SUMMARY:
This research study will assess the real-world effectiveness of Facebook advertising as a strategy to reach women of reproductive age who are at risk of unintended pregnancy with a brief educational intervention about emergency contraception (EC).

DETAILED DESCRIPTION:
This research study will assess the real-world effectiveness of Facebook advertising as a strategy to reach women of reproductive age who are at risk of unintended pregnancy with a brief educational intervention about emergency contraception (EC). The investigators will assess whether a video or website link has superior reach, engagement, and return on investment (measured as cost per click) through a Facebook ad campaign. The investigators will also ensure that both modalities of consumer engagement (website and video) are efficacious at ensuring adequate and improved knowledge of emergency contraception through a laboratory-environment trial.

ELIGIBILITY:
Inclusion Criteria:

* Women
* 18 to 29 years old
* Living or seeking care in or around Boston, MA
* Able to participate in an in-person visit at Planned Parenthood League of Massachusetts (PPLM) Boston Health Center
* English fluency
* Have at least one social media account (i.e. Facebook, Instagram, Twitter, Pinterest, YouTube, Snapchat)
* Endorse using social media at least once a week

Exclusion Criteria:

* PPLM staff
* Currently or ever employed in the reproductive health field
* Currently using long-acting reversible contraception (LARC)
* History of permanent sterilization (by participant or sexual partner)
* Previous participation in the study

Ages: 18 Years to 29 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 150 (Actual)
Dates: Start 2019-01-15 (Actual); Primary Completion 2019-06-07 (Actual); Study Completion 2019-06-07 (Actual)

PRIMARY OUTCOMES:
Emergency contraception knowledge (binary) | Immediately after intervention
  This outcome is a binary outcome that reflects a participant's ability to correctly identify an emergency contraceptive method, when to use it, and how to access it

SECONDARY OUTCOMES:
Copper IUD as emergency contraception knowledge | Immediately after intervention
  This outcome is a binary outcomes that reflects a participant's ability to correctly identify the copper IUD as emergency contraception, when to use it, and how to access it.
Levonorgestrel pill as emergency contraception knowledge | Immediately after intervention
  This outcome is a binary outcomes that reflects a participant's ability to correctly identify the levonorgestrel pill as emergency contraception, when to use it, and how to access it.
Ulipristal pill as emergency contraception knowledge | Immediately after intervention
  This outcome is a binary outcomes that reflects a participant's ability to correctly identify the ulipristal pill as emergency contraception, when to use it, and how to access it.
Emergency contraception knowledge (continuous) | Immediately after intervention
  This outcome reflects the participant's overall knowledge of emergency contraception after the website or video intervention, as measured by the proportion of questions they get correct on the survey
Change in emergency contraception knowledge pre- and post-intervention | Immediately before and immediately after intervention
  This outcome reflects the participant's change in knowledge of emergency contraception before and after the website or video intervention, as measured by the proportion of questions they get correct on the survey.
Likelihood of using emergency contraception pre- and post-intervention | Immediately before and immediately after intervention
  This outcome reflects the participant's likelihood of using emergency contraception both before and after the intervention, as measured on a 6 point likert scale (I would definitely use it, Very likely, Somewhat likely, Somewhat unlikely, Very unlikely, I definitely would NOT use it)

CONTACTS AND LOCATIONS:
Overall Officials: Principal Investigator, MD, Principal Investigator — Planned Parenthood League of Massachusetts
Locations (1):
- PPLM, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No